CLINICAL TRIAL: NCT01647490
Title: Right Ventricular Lead Placement in a Pacemaker Population: Evaluation of Apical and Alternative Position - Right Pace Study
Brief Title: Right Ventricular Lead Placement in a Pacemaker Population: Evaluation of Apical and Alternative Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Santa Maria di Loreto Mare (Other)
Responsible Party: Principal Investigator, Carmine Muto, Electrophysiology and Pacing Unit Director, Ospedale Santa Maria di Loreto Mare
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LM-003
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Bradycardia; Heart Block; Sick Sinus Syndrome
MeSH Terms: conditions — Bradycardia; Heart Block; Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right Ventricular Apex (RVA) (Active Comparator): In the RVA group the right ventricular pacing lead will be implanted in the apex region of the right ventricle
  Interventions: Procedure: Permanent Cardiac Pacemaker Implantation
- Right Ventricular Septum (RVS) (Experimental): In the RVS group the right ventricular pacing lead will be implanted in the septal region (mid septum) of the right ventricle
  Interventions: Procedure: Permanent Cardiac Pacemaker Implantation

INTERVENTIONS:
Procedure: Permanent Cardiac Pacemaker Implantation

SUMMARY:
This study is a long-term, prospective, and controlled evaluation of the mechanical dyssynchrony induced by right ventricular apical pacing, both in acute (spontaneous and stimulated) and chronic (12 and 24 months); the study also evaluates the benefit of an alternative pacing site through measures of dyssynchrony in acute and chronic.

DETAILED DESCRIPTION:
Permanent cardiac pacing plays an important role in cardiac disease management. Since early studies on right ventricular pacing, apex has been the preferred implant site for transvenous endocardial ventricular leads for several reasons: ease of placement, lead stability as well as the design characteristics of the electrode and the fixation system.

It is now also accepted, however, that right ventricle pacing causes a long term deterioration of left ventricular function through complex effects, both at the structural level of the heart wall and at the hemodynamic level in left ventricular load conditions. It is possible that this deterioration is due to a dyssynchrony of contraction induced by pacing at the right ventricular apex. Some authors suggest to pace the right ventricle at alternative sites, i.e. the medium septum (RVS) region, to guarantee a more physiological activation pattern, especially in patients expected to receive high pacing percentages.

However, unequivocal evidences that stimulation of the right ventricular septum is more physiological than the apical pacing are still missing.

Nonetheless, it should be noted that, although a number of studies refer to RV septum as the alternative site for pacing , poor attention has been paid to the unambiguous definition of RV septum region itself. A clear definition and a proper evaluation of the alternative site is therefore important.

Furthermore, from a procedural point of view, it has been demonstrated that acute and chronic electrical performances of the leads positioned at alternative sites, in particular in the region of mid septum, are equivalent to those of the leads positioned at the apical site.

The purpose of this study is to perform a comprehensive assessment of the electrical and mechanical measures obtained by pacing standard RV site (Right ventricular apex, RVA) and alternative RV site (right ventricular septum, RVS). Specifically, the two pacing sites will be compared in terms of electrical dyssynchrony, as assessed by ECG criteria, and in terms of mechanical dyssynchrony, as assessed by echocardiographic criteria.

The primary end point of the study is defined through the evaluation of dyssynchrony measured both in spontaneous rhythm (Vs) and paced rhythm (Vp). The delay between the time to peak systolic velocity of the septum and the LV free wall will be used to define the degree of dyssynchrony; this measurement will be obtained by TDI echocardiographic technique.

Patients will receive any commercially available dual-chamber implantable pacemakers, according to current standard indications. At the end of the implantation and at follow-up visits (12 and 24 months) device programming will follow the clinical practice of the center.

ELIGIBILITY:
Inclusion Criteria:

* indication for a dual chambers cardiac pacemaker device (DDD/DR) according to current guidelines
* Patients who are able to understand and sign an informed written consent
* Patients who will conduct the follow-up in the center for at least 24 months
* Patients age ≥ 18

Exclusion Criteria:

* Patients with chronic atrial fibrillation or atrial arrhythmias not controlled within 90 days before enrollment
* Pre-existing permanent cardiac pacemaker (PM), defibrillator (ICD) or cardiac resynchronization therapy device (CRT)
* Unplanned or emergency access to the hospital and / or inability to measure the dyssynchrony for the absence of spontaneous rhythm
* Patients participating in other studies that clearly impact the clinical practice of the center or whose protocol would conflict or affect the outcome of this study
* Patient not expected to survive for the duration of the study follow-up due to co-morbid medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
LV dyssynchrony as measured by Electromechanical delay (EMD | 2 weeks
  The primary outcome measure of this study is to compare the effect of RV Septal (RVS) versus RV Apical (RVA) pacing as measured by echocardiographic/Doppler Index

SECONDARY OUTCOMES:
Number of heart failure-related hospitalization | 24 months
  To compare the rate of heart failure-related hospitalization between RVS versus RVA pacing
Right ventricular lead and total implant procedure time, fluoroscopy time | Implant
  To compare the procedural time of RVS versus RVA pacing
Change from baseline in R wave in 12-lead ECG | 24 months
  To investigate the relationship between the ECG characteristics at baseline and response to cardiac pacing (as measured by echocardiography as defined in primary outcome measure) at implant and 24 months
Absolute change in LVEF | 24 months
  To evaluate the Left ventricular diastolic and systolic function as measured by Echocardiographic response of absolute change in LVEF
LV dyssynchrony as measured by Electromechanical delay (EMD) | 24 months
  The secondary outcome measure of this study is to compare the effect of RVS versus RVA pacing as measured by echocardiographic/Doppler Index. This extends to 24 months the results obtained with the primary objective at 2 weeks
Symptoms and quality of life scores | 24 months
  To investigate the relationship between the right ventricular lead position and response to cardiac pacing in terms of symptoms and quality of life scores as measured by short form (SF)-12 scores

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Muto, MD, Study Chair — Ospedale Santa Maria di Loreto Mare; Valeria Calvi, MD, Study Chair — Azienda Ospedaliero Universitaria "Vittorio Emanuele" - Ferrarotto
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria "Vittorio Emanuele", Catania
  - Ospedale Santa Maria di Loreto Mare, Naples

REFERENCES:
- [Derived] Muto C, Calvi V, Botto GL, Pecora D, Porcelli D, Costa A, Ciaramitaro G, Airo Farulla R, Rago A, Calvanese R, Baratto MT, Reggiani A, Giammaria M, Patane S, Campari M, Valsecchi S, Maglia G. Chronic Apical and Nonapical Right Ventricular Pacing in Patients with High-Grade Atrioventricular Block: Results of the Right Pace Study. Biomed Res Int. 2018 May 22;2018:1404659. doi: 10.1155/2018/1404659. eCollection 2018. PMID 29951525
- [Derived] Muto C, Calvi V, Botto GL, Pecora D, Ciaramitaro G, Valsecchi S, Malacrida M, Maglia G. Is there a right place to pace the right ventricle? Evaluation of apical and septal positions in a pacemaker population: study protocol for a prospective intervention-control trial. Contemp Clin Trials. 2014 Nov;39(2):320-6. doi: 10.1016/j.cct.2014.10.006. Epub 2014 Oct 22. PMID 25465496